CLINICAL TRIAL: NCT02658526
Title: Role of Anesthesia / Surgery on Cognitive Function in Child
Brief Title: Cognitive Changes in Childs After Anesthesia / Surgery
Status: Withdrawn | Type: Observational
Why Stopped: Problems in organization
Sponsor: Konstanze Plaschke (Other)
Responsible Party: Sponsor-Investigator, Konstanze Plaschke, Prof., Heidelberg University
Organization: Heidelberg University (Other)
Other Study IDs: S-086/2014
Record Dates: First submitted 2015-12-08; First posted 2016-01-20 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Behavioral
Keywords: cognition; anesthesia; surgery; stress; child
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- control: children without anesthesia / surgery
- anesthesia: children with anesthesia for diagnostic reason
  Interventions: Behavioral: anesthesia - surgery
- surgery: children with anesthesia / surgery
  Interventions: Behavioral: anesthesia - surgery

INTERVENTIONS:
Behavioral: anesthesia - surgery
  Groups: anesthesia; surgery

SUMMARY:
The role of surgical stress and anesthesia is unknown in the early childhood. In vitro and animal studies showed a risk for treatment with anesthesia in the developmental brain. Furthermore, stress is also an important risk factor for cognitive impairment. Therefore, the investigators want to investigate in a clinical prospective cohort study the role anesthesia and surgery on different cognitive parameters and self-controling mechanisms in children under 3 years.

DETAILED DESCRIPTION:
In order to investigate the role of anesthesia and / or surgery on cognitive abilities the investigators want to perform a prospective cohort study in children under 3 years. Three groups should be compared: i) control without anesthesia / surgery, ii) children with only anesthesia, and iii) children with both surgery and anesthesia. All children will be investigate before and after intervention. Different behavioral scales will be used for detailed cognitive abilities and self-regulatory skills.

ELIGIBILITY:
Inclusion Criteria:

* Age 9 month to 3 years with or without anesthesia / surgery

Exclusion Criteria:

* Psychiatrical, neurological, oncological diseases

Ages: 9 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Cohort study - children <3 years
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Global cognitive abilities | 4-6 weeks
  Bayley Scale
Global cognitive abilities | 4-6 weeks
  MONDEY (Milestone of Normal Development in Early Years) Scale
Global cognitive abilities | 4-6 weeks
  Assessment of temperament with the Infant Behavior Questionnaire Revised (IBQ-R) questionnaire
Global cognitive abilities | 4-6 weeks
  Early Childhood Behavior Questionnaire (ECBQ) questionnaire

SECONDARY OUTCOMES:
surgery-associated data | 1 - 3 days
  reason of surgery
surgery-associated data | 1 day
  date of birth
surgery-associated data | 1 day
  length of surgery (h:min)
surgery-associated data | 1 day
  kind and quantity of anesthesia and medication (number)
surgery-associated data | 1 day
  Age (month)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Heidelberg, Department of Anesthesiology, Heidelberg Medical School, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No